CLINICAL TRIAL: NCT01762748
Title: Effect of Saccharomyces Boulardii in Patients in the Waiting List for Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Juliana Costa Liboredo, Fellow PhD degree, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETIC 0609.0.203.000-09
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Liver Cirrhosis
Keywords: Probiotic; liver; transplant; permeability
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S. boulardii 200mg (Floratil®) (Experimental): The patients received S. boulardii every 8h during 30 days as an oral capsule formulation which contained 200 mg lyophilized S. boulardii-17 (Floratil®).
  The patients enrolled in the study were evaluated immediately before the beginning of treatment, after a thirty-day period of treatment with probiotic and at the end of the second study month (after a thirty-day period without treatment with probiotic).
  Interventions: Drug: Saccharomyces boulardii

INTERVENTIONS:
Drug: Saccharomyces boulardii — Oral capsule with 200 mg lyophilized S. boulardii-17 (about 4x108 cells), 6 mg sucrose and 2.4 mg magnesium stearate (Floratil®).
  Other Names: Floratil

SUMMARY:
The purpose of this study is to evaluate the effect of Saccharomyces boulardii in patients in the waiting list for liver transplant.

DETAILED DESCRIPTION:
Increased intestinal permeability are related to the major complications of liver cirrhosis. The administration of probiotics has been suggested to improve the barrier function of the mucosa and consequently avoid the complications of the disease. The objective of this study was to evaluate the effect of Saccharomyces boulardii in patients in the waiting list for liver transplant.

Eighteen patients were treated with Saccharomyces boulardii. Intestinal permeability (lactulose/mannitol ratio) and laboratory parameters were evaluated immediately before the beginning of treatment, after a thirty-day period of treatment with probiotic and at the end of the second study month (after a thirty-day period without treatment with probiotic). Twenty healthy volunteers were also submitted for the intestinal permeability test.

ELIGIBILITY:
Inclusion Criteria:

* patients in the waiting list for liver transplant with viral, alcoholic or cryptogenic cirrhosis

Exclusion Criteria:

* patients younger than 18 years or older than 65 years.
* patients with renal failure, congestive heart failure, nephrotic syndrome, diabetes and thyroid diseases that interfered with absorption, flux of water and solutes and intestinal motility, in order to avoid interference with the intestinal permeability tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability | Change from intestinal permeability at two months
  Intestinal permeability test was conducted at the lactulose and mannitol excretion

SECONDARY OUTCOMES:
Effect of Saccharomyces boulardii on laboratory parameters | Change from laboratory parameters in two months
Number of participants with adverse effect | Adverse effect in two months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel Correia, PhD, Study Chair — Federal University of Minas Gerais; Juliana Liboredo, PhD degree, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Alfa Institute of Gastroenterology - Transplant Outpatient Clinic at Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil